CLINICAL TRIAL: NCT03690011
Title: Cell Therapy for High Risk T-cell Malignancies Using CD7-Specific CAR Expressed on Non-Edited T Cells (CRIMSON-NE)
Brief Title: Cell Therapy for High Risk T-Cell Malignancies Using CD7-Specific CAR Expressed On Autologous T Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Leukemia and Lymphoma Society (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, LaQuisa Hill, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43761 - CRIMSON NE
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: T-cell Acute Lymphoblastic Lymphoma; T-non-Hodgkin Lymphoma; T-cell Acute Lymphoblastic Leukemia
Keywords: Autologous CAR T cells; T-cell acute lymphoblastic lymphoma; T-non-Hodgkin lymphoma; T-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD7.CAR/28zeta CAR T Cells (Experimental): Four dose levels will be evaluated. The T cells will be administered following lymphodepleting chemotherapy with cyclophosphamide and fludarabine.
  Interventions: Genetic: CD7.CAR/28zeta CAR T cells

INTERVENTIONS:
Genetic: CD7.CAR/28zeta CAR T cells — Three dose levels will be evaluated:
  * Dose level one: 1×10^7 cells/m^2
  * Dose level two: 3×10^7 cells/m^2
  * Dose level three: 5x10^7 cells/m^2
  * Dose level four: 1×10^8 cells/m^2

SUMMARY:
Patients eligible for this study have a type of blood cancer called T-cell leukemia or lymphoma (lymph gland cancer).

The body has different ways of fighting infection and disease. This study combines two different ways of fighting disease with antibodies and T cells. Antibodies are types of proteins that protect the body from bacterial and other diseases. T cells, or T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. Both antibodies and T cells have been used to treat cancer; they have shown promise, but have not been strong enough to cure most patients.

T cells can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study is called anti-CD7. This antibody sticks to T-cell leukemia or lymphoma cells because of a substance on the outside of these cells called CD7. CD7 antibodies have been used to treat people with T-cell leukemia and lymphoma. For this study, anti-CD7 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor.

In the laboratory, investigators have also found that T cells work better if they also add proteins that stimulate T cells, such as one called CD28. Adding the CD28 makes the cells grow better and last longer in the body, thus giving the cells a better chance of killing the leukemia or lymphoma cells.

In this study, investigators attach the CD7 chimeric receptor with CD28 added to it to T cells. Investigators will then test how long the cells last. These CD7 chimeric receptor T cells with CD28 are investigational products not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
To make the T cells, the investigators will take the patient's blood and stimulate it with growth factors to make the T cells grow. To get the CD7 antibody and CD28 to attach to the surface of the T cell, investigators will insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps investigators find the T cells in the patient's blood after investigators inject them. This virus also helps the investigators find the T cells in your blood after they are injected. To ensure the T cells grow well in the lab, the investigators adds small amounts of medications that are often used to treat patients with cancer or other illnesses. These medications are washed off of the cells prior to injecting them into your body. Because patients will have received cells with a new gene in them, patients will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. If patients cannot visit the clinic, they may be contacted by the research coordinator or physician.

When patients enroll on this study, they will be assigned a dose of CD7 chimeric receptor-T cells. Several studies suggest that the infused T cells need room to be able to proliferate (grow) and accomplish their functions and that this may not happen if there are too many other T cells in blood. Because of that, patients will receive two chemotherapy medications prior to receiving the CD7 chimeric receptor-T cells. One medication is called cyclophosphamide and the other fludarabine. Patients will receive 3 daily doses of each drug, ending at least one day before they receive the chimeric receptor-T cells. These drugs will decrease the numbers of the patients own T cells before investigators infuse the CD7 chimeric receptor T cells and also will help decrease the number of other cells that may interfere with the chimeric receptor-T cells working well. Although investigators do not expect any effect on tumors with the doses that patients will receive, these drugs are part of many regimens that are used to treat leukemia or lymphoma. Investigators prefer that patients do not receive other chemotherapy or treatments for your cancer until 4 weeks after cell infusion but patients can do so if their doctors thinks it is medically necessary.

Patients will be given an injection of cells into the vein through an IV at the assigned dose. Before patients receive the injection, they will be given a dose of Benadryl and Tylenol. The injection will take about 1-10 minutes. Investigators will follow patients in the clinic after the injection at least 3 hours post infusion, and they will have to remain locally for at least 3 weeks after the infusion. If patients experience any side effects (see section on risks below), they may have to be hospitalized for evaluation and management. If after a 4-6 week evaluation period after a patient's infusion and s/he has achieved a complete response (measured by bone marrow or radiology scans), the patient's primary oncology doctors may decide s/he should proceed to bone marrow transplant, at which time s/he will be removed from the treatment portion of the study.

The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

MEDICAL TESTS BEFORE TREATMENT

Before being treated, patients will receive a series of standard medical tests:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the patient's tumor by scans and/or bone marrow studies
* Testing of patient's blood for certain viral infections
* An ultrasound of patient's heart to make sure his/her heart function is appropriate for the study if you have not had one recently

MEDICAL TESTS DURING AND AFTER TREATMENT:

Patients will receive standard medical tests when they are getting the infusion and after:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the patient's tumor by scans and/or bone marrow studies 4-6 weeks after the infusion

To learn more about the way the CD7 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn. The total amount on any day is about 10 teaspoons (50 mL) or no more than 3 mL per 2.2 pounds body weight in children. This volume is considered safe but may be decreased if patients are anemic. This blood may be drawn from a central line if one is available. Blood will be taken before patients start the chemotherapy a few days prior to the cell infusion. On the day patients receive the cells, blood will be taken before the cells are given and several hours afterwards. Other blood will be drawn one week after the infusion, 2 weeks, 3 weeks, 4 weeks, 6 weeks and 8 weeks after the infusion, at 3 months, at 6 months, at 9 months, at 1 year, every 6 months for 4 years, then yearly for a total of 15 years. The total blood drawn during a patient's participation in this study will not exceed 280 teaspoons.

ELIGIBILITY:
Procurement Inclusion Criteria:

Referred patients will initially be consented for procurement of blood for generation of the transduced ATL. Eligibility criteria at this stage include:

1. Diagnosis of recurrent or refractory T-cell acute lymphoblastic leukemia (T-ALL), T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher) or other cutaneous T-cell lymphomas

AND

1. suitable for allogeneic hematopoietic stem cell transplant (HSCT)
2. with a suitable donor identified by a FACT accredited transplant center
3. willing to proceed to transplant if the CD7.CAR treatment induces complete remission and the patient/donor remain suitable candidates

Using NMDP donor assessment criteria, suitability is defined as "during the search process, a donor is medically fit to proceed to the next step- whether high-resolution or confirmatory HLA testing OR donor work-up." Documentation of suitability (including above criteria) will be confirmed by the investigator prior to treatment.

* For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.

  2. CD7-positive tumor (≥20% CD7 positive blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory).

  3. Age </=75 years old.. NOTE: The first three (3) patients treated on the study must be adults (>/=18 yrs of age).

  4. Hgb ≥ 7.0 (can be transfused)

  5. Life expectancy greater than 12 weeks

  6. If pheresis required to collect blood:
  * Cr < 1.5 upper limit normal
  * AST < 5 × upper limit normal
  * PT and APTT <1.5 × upper limit normal

    7. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Procurement Exclusion Criteria:

1. Active infection requiring antibiotics.
2. Active infection with HIV
3. History of other cancer (except non-melanoma skin cancer or in situ breast cancer or cervix cancer) unless the tumor was successfully treated with curative intent at least 2 years before trial entry.

Treatment Inclusion Criteria:

1. Diagnosis of recurrent or refractory T-cell acute lymphoblastic leukemia (T-ALL),T-cell acute lymphoblastic lymphoma (T-LLy), or T-non-Hodgkin lymphoma (T-NHL, including Angioimmunoblastic T-cell lymphoma (AITL), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Peripheral T-cell lymphoma (PTCL) NOS, Anaplastic large cell lymphoma (ALCL), Adult T-cell leukemia/lymphoma, T cell prolymphocytic leukemia with symptomatic disease, Extranodal NK/T cell lymphoma, Mycosis fungoides/ Sezary Syndrome Stage IIB or higher) or other cutaneous T-cell lymphomas

AND

1) suitable for allogeneic hematopoietic stem cell transplant (HSCT) 2) with a suitable donor identified by a FACT accredited transplant center 3) willing to proceed to transplant if the CD7.CAR treatment induces complete remission and the patient/donor remain suitable candidates

Using NMDP donor assessment criteria, suitability is defined as "during the search process, a donor is medically fit to proceed to the next step- whether high-resolution or confirmatory HLA testing OR donor work-up." Documentation of suitability (including above criteria) will be confirmed by the investigator prior to treatment.

* For T-NHL subjects, eligibility will be confined to disease stages where allogeneic HSCT is indicated.

  2. CD7-positive tumor (≥20% CD7+ blasts by flow cytometry or immunohistochemistry (tissue) assessed in a CLIA certified Flow Cytometry/Pathology laboratory.

  3. Age </=75 years old. NOTE: The first three (3) patients treated on the study must be adults (>/=18 yrs of age).

  4. Bilirubin less than 3 times the upper limit of normal.

  5. AST less than 5 times the upper limit of normal.

  6. Estimated GFR ≥ 50 mL/min.

  7. Pulse oximetry of > 90% on room air

  8. Karnofsky or Lansky score of ≥ 60.

  9. Recovered from acute toxic effects of prior chemotherapy at least one week before entering this study.

  10. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.

  11. Informed consent explained to, understood by, and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Exclusion Criteria:

1. Currently receiving any investigational agents or having received any tumor vaccines within the previous 6 weeks.
2. History of hypersensitivity reactions to murine protein-containing products.
3. Pregnant or lactating.
4. Tumor in a location where enlargement could cause airway obstruction (per investigator discretion).
5. Clinically significant viral infection or uncontrolled viral reactivation of EBV, CMV, Adv, BK-virus, or HHV-6.
6. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF≤30% or LVEF≤50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment).
7. CNS abnormalities: Presence of CNS-3 disease defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm3 (unless negative by the Steinherz/Bleyer algorithm); Presence of any CNS disorder such as an uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage within the past 12 months, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2040-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | 4 weeks
  To evaluate the safety of escalating doses of autologous peripheral blood T lymphocytes (ATLs) genetically modified to express chimeric antigen receptors (CAR) targeting the CD7 molecule (CD7.CAR) in combination with lymphodepletion in patients with relapsed/refractory T-cell malignancies.

SECONDARY OUTCOMES:
Overall Response Rate | 4 weeks
  To measure the anti-tumor effects of CD7.CAR-ATLs in patients with T-cell leukemia or lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Rayne Rouce, MD, Principal Investigator — Pediatrics, Baylor College of Medicine; LaQuisa Hill, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Velasquez MP. Allogeneic CD7-CAR T cells to bridge the gap? Transplant Cell Ther. 2023 Mar;29(3):139-140. doi: 10.1016/j.jtct.2023.02.006. No abstract available. PMID 36858787
- [Derived] Watanabe N, Mo F, Zheng R, Ma R, Bray VC, van Leeuwen DG, Sritabal-Ramirez J, Hu H, Wang S, Mehta B, Srinivasan M, Scherer LD, Zhang H, Thakkar SG, Hill LC, Heslop HE, Cheng C, Brenner MK, Mamonkin M. Feasibility and preclinical efficacy of CD7-unedited CD7 CAR T cells for T cell malignancies. Mol Ther. 2023 Jan 4;31(1):24-34. doi: 10.1016/j.ymthe.2022.09.003. Epub 2022 Sep 9. PMID 36086817